CLINICAL TRIAL: NCT04374019
Title: Randomized, Multi-arm Phase II Trial of Novel Agents for Treatment of High-risk COVID-19 Positive Patients
Brief Title: Novel Agents for Treatment of High-risk COVID-19 Positive Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual,
Sponsor: Susanne Arnold (Other)
Responsible Party: Sponsor-Investigator, Susanne Arnold, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20-COVID-01-PMC
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Results first posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: COVID; Sars-CoV2
Keywords: high-risk
MeSH Terms: interventions — Ivermectin; camostat; Artesunate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Arm C: Ivermectin (Experimental): Ivermectin
  Interventions: Drug: Ivermectin
- Arm D: Camostat Mesilate (Experimental): Camostat Mesilate
  Interventions: Drug: Camostat Mesilate
- Arm E: Artemesia annua (Experimental): Artemesia annua tea or coffee
  Interventions: Dietary Supplement: Artemesia annua
- Arm F: Artesunate (Experimental): Artesunate
  Interventions: Drug: Artesunate

INTERVENTIONS:
Drug: Ivermectin — Ivermectin:
  Days 1-2: Weight < 75kg: 4 tabs (12 mg total daily dose) Days 1-2: Weight > 75kg: 5 tabs (15 mg total daily dose)
  Arms: Arm C: Ivermectin
Drug: Camostat Mesilate — Days 1-14: 2 tab TID after a meal (600 mg total daily dose)
  Arms: Arm D: Camostat Mesilate
Dietary Supplement: Artemesia annua — Days 1-14: tea or coffee pod TID (1350 mg total daily dose)
  Arms: Arm E: Artemesia annua
Drug: Artesunate — Days 1-14:
  Arms: Arm F: Artesunate

SUMMARY:
This is a multi-arm, phase II trial for rapid efficacy and toxicity assessment of multiple therapies immediately after COVID19 positive testing in high-risk individuals. Therapies include stand-alone or combination treatment with hydroxychloroquine, azithromycin, ivermectin, or camostat mesilate, artemesia annua. The hypothesis of this study is that the addition of agents that inhibit viral entry or replication of SARS-CoV-2 virus replication in will be devoid of additional moderate to severe toxicities, will prevent clinical deterioration, and will improve viral clearance in high risk individuals.

DETAILED DESCRIPTION:
Coronavirus Disease 2019 (COVID-19) is a highly contagious disease, caused by a novel enveloped RNA beta-coronavirus, also known as severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2). The first case of this unprecedented outbreak "pneumonia of unknown etiology" was reported in Wuhan City, Hubei Province, China on December 8th, 2019 and reported to the World Health Organization (WHO) on December 31st, 2019. WHO declared a COVID-19 global emergency on January 30, 2020, and then categorized the outbreak as a pandemic on March 11, 2020. As of April 22, 2020, more than 2,628,894 confirmed cases of COVID-19 worldwide and 182,740 people globally have died from COVID-19 since it emerged in China, according to the data from Johns Hopkins University.

While the majority of patients with COVID-19 develop mild or uncomplicated illness, approximately 20-30% of hospitalized patients have required intensive care support and 5% of those have multi-organ failure or shock. The case fatality rate ranges from 1 to 4% and it is higher among those with pre-existing comorbid conditions such as cardiovascular disease, diabetes mellitus, obesity, chronic respiratory disease, hypertension and cancer. The vast majority of patients present with fever (83-99%), cough (59-82%), fatigue (44-70%), anorexia (40-84%), shortness of breath (31-40%), sputum production (28-33%), myalgias (11-35%). Less than 10% of patients will present with headache, confusion, rhinorrhea, sore throat, hemoptysis, vomiting, or diarrhea. Anosmia or ageusia proceeding the onset of respiratory symptoms has been anecdotally reported.

To date, treatments for COVID-19 in high risks individuals remain experimental and therapeutic strategies to deal with the infection are at best supportive, with prevention aimed at reducing transmission in the community as the best weapon. No proven therapies have been demonstrated to prevent the progression of COVID-19 to severe illness and this is a critical unmet need for high-risk individuals and warrants study. Recently, the Infectious Disease Society of America has made recommendations for the treatment of patients with COVID-19, focusing on inpatient care, and recommending randomized trials where possible as the best step to improve treatment outcomes and to increase our understanding of this coronavirus pandemic. Discoveries in this area may inform clinicians on effective treatment for low-risk individuals who progress to severe illness, as well.

ELIGIBILITY:
Inclusion Criteria

* Age ≥18 years
* Laboratory-confirmed SARS-CoV-2 infection within the past 7 days or the presence of symptoms or physical examination signs providing high probability of COVID-19 disease
* Patients must have adequate organ and marrow function measured within the last 6 months
* Subjects must have at least one of the following high-risk features for clinical deterioration:

  * Hypertension
  * Diabetes Mellitus
  * Moderate to severe Chronic Obstructive Pulmonary Disease, Emphysema, Cystic Fibrosis, or Asthma
  * Cancer patients who have received any immunosuppressive drugs within a year from enrollment
  * Sickle Cell disease or thalessemia
  * Age > or = 50
  * BMI > or = 30
  * Living in a nursing home or long-term facility
  * Underlying serious heart condition as determined by the treating physician
  * Immunocompromised subject as defined by the treating physician or COVID-19 Telehealth Treatment Team

Exclusion Criteria

* Severe or life threating COVID
* Weight less than 45 kg.
* Pregnant or breast-feeding females
* Subjects on dialysis or with creatinine clearance < 45 ml/min
* Existing DMID Toxicity Scale for Determining Severity of Adverse Events grade 3 or greater hepatic failure
* Previously documented moderate or severe retinopathy or macular degeneration
* Uncontrolled Seizure disorder
* Prolonged QT, defined as QTc ≥470 milliseconds for men and as QTc ≥480 for women using Bazett's formula
* Known allergy to artesunate, artemisia annua, hydroxychloroquine, macrolides, 4-aminoquinolines, camostat mesilate, or other agents to be used in the trial.
* Currently receiving any study medications for other indications
* Concurrent use of medication that would cause drug-drug interactions
* Patients with psychiatric illness/social situations that would limit compliance

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2022-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Arnold, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period 5/1/2020 to 11/23/2020; Study on hold for most of 2021, terminated in early 2022 due to low accrual
Groups:
- Arm A - Hydrozychloroquine: Hydroxychloroquine 600 mg daily Days 1-14
- Arm B - Hydroxychloroquine + Azithromycin: Hydroxychloroquine 600 mg daily Days 1-14
  + Azithromycin 500 mg Day 1; 250 mg daily Days 2-5
- Arm C - Ivermectin: Ivermectin 12-15- mg (weight based) on Day 1 and 2
- Arm D - Camostat: Camostat 200mg TID Days 1-14
Period: Overall Study
Arm/Group | Arm A - Hydrozychloroquine | Arm B - Hydroxychloroquine + Azithromycin | Arm C - Ivermectin | Arm D - Camostat
Started | 1 | 1 | 6 | 5
Completed | 1 | 1 | 5 | 5
Not Completed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Hydroxychloroquine
- Arm B: Hydroxychloroquine + Azithromycin
- Arm C: Ivermectin
  Ivermectin: Ivermectin:
  Days 1-2: Weight < 75kg: 4 tabs (12 mg total daily dose) Days 1-2: Weight > 75kg: 5 tabs (15 mg total daily dose)
- Arm D: Camostat Mesilate
  Camostat Mesilate: Days 1-14: 2 tab TID after a meal (600 mg total daily dose)
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Arm D | Total
Number analyzed (Participants) | 1 | 1 | 6 | 5 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 5 | 3 | 10
  >=65 years | 0 | 0 | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 4 | 8
  Male | 0 | 1 | 3 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 6 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 6 | 5 | 13
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — COVID-19 positive by PCR
  participants
    United States | 1 | 1 | 6 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Clinical Deterioration
Description: Number of patients experiencing clinical deterioration. Clinical deterioration is defined as a less than a 2-point change from the initial COVID 7-Point Ordinal Outcomes Scale within 14 days from the study start. This scale ranges from 1-7. Lower scores indicate worse outcomes (death); higher scores indicate fewer symptoms and better outcomes.
Time Frame: 14 days
Population: 1 subject was inevaluable in Arm C. No subjects clinically deteriorated as defned above
Measure: Count of Participants; unit: Participants
Groups:
- Arm C: Ivermectin
- Arm D: Camostat
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 1 | 1 | 5 | 5
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Change in Viral Load
Description: The change in (clearance of) viral RNA will be measured by PCR testing at days 1, 14, 28, and 40 days.
Time Frame: 40 days
Population: study terminated due to low accrual, no subjects analyzed for this outcome.
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Rate of Organ Failure
Description: Number of patients that experienced severe respiratory or other organ failure.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 1 | 1 | 5 | 5
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Progression to ICU Care or Ventilation
Description: Percentage of patients requiring ICU admission or ventilation.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 1 | 1 | 5 | 5
Participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants Who Had a Change in Clinical Status Measured by Decrease in COVID 7-point Ordinal Scale
Description: Number of participants who died or had greater than a 2-point decrease in COVID 7-Point Ordinal Outcomes Scale from Day to Day 14.
  COVID 7-point ordinal outcomes scale:
  1. Death
  2. Hospitalized on invasive mechanical ventilation or ECMO
  3. Hospitalized on non-invasive ventilation or high flow nasal cannula
  4. Hospitalized on supplemental oxygen
  5. Hospitalized not on supplemental oxygen
  6. Not hospitalized with limitation in activity (continued symptoms)
  7. Not hospitalized without limitation in activity (no symptoms)
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 1 | 1 | 5 | 5
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Mortality
Description: Percentage of patients who have died by day 14.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 1 | 1 | 5 | 5
Participants | 0 | 0 | 0 | 0

7. Secondary Outcome: Rate of Severe Adverse Events
Description: Percentage of patients experiencing severe adverse events, defined as grade 3 non-hematologic or greater by DMID Toxicity Scale for Determining Severity of Adverse Events.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 1 | 1 | 5 | 5
Participants | 1 | 0 | 1 | 0

8. Secondary Outcome: Number of Patients That Required Oxygen Supplementation
Description: Number of patients that required oxygen supplementation during study treatment Days 1-28
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 1 | 1 | 5 | 5
Participants | 1 | 1 | 1 | 1

9. Secondary Outcome: Number of Patients That Required Mechanical Ventilation
Description: Number of patients that required mechanical ventilation during the study period. Days 1-28
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 1 | 1 | 5 | 5
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Patients Who Required Vasopressors
Description: Number of patients who required vasopressor treatment Days 1 to 28
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 1 | 1 | 5 | 5
Participants | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Patients Who Required ICU Services
Description: Number of patients who required ICU services during study treatment Days 1-28.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 1 | 1 | 5 | 5
Participants | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Patients That Required Hospitalization
Description: Number of patients that required hospitalization during study treatment
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 1 | 1 | 5 | 5
Participants | 0 | 0 | 4 | 4

13. Secondary Outcome: Heart Function
Description: Proportion of patients with significant changes in ECG findings, including heart rate, ECG intervals (PR, QTcB, QTcF), conduction changes, or abnormalities including severe QTc prolongation of > 500 ms.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 1 | 1 | 5 | 5
Participants | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: AEs were collected from study entry until Day 28.
Arm/Group | Arm A | Arm B | Arm C | Arm D
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 1/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 1/5 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=1) | Arm B (N=1) | Arm C (N=5) | Arm D (N=5)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — grade 4 anemia, unrelated to HCQ, but related to underlying malignancy
supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — SVT possibly due to ivermectin, resolved
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=1) | Arm B (N=1) | Arm C (N=5) | Arm D (N=5)
mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — mucositis oral, grade 2, definitely related
GERD (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — grade 1, possibly related
tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — grade 1 tinnitus, possibly related

LIMITATIONS AND CAVEATS:
Thsi study was closed to accrual due to slow accrual rate. No conclusions on efficacy can be made due to a lack of statistical power in each arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT04374019/Prot_SAP_000.pdf